CLINICAL TRIAL: NCT04006275
Title: Comparing SonoVue With Sonazoid in the Performance of Contrast Enhanced Ultrasound The Liver Imaging Reporting and Data System (CEUS-LIRADS) in Diagosing HCC: a Prospective Blind Study
Brief Title: Comparing SonoVue With Sonazoid Using CEUS-LIRADS in HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 研2019-073
Record Dates: First submitted 2019-06-25; First posted 2019-07-05 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
Keywords: Hepatocellular Carcinoma; cirhossi; Contrast-enhanced ultrasound; LI-RADS
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis | interventions — contrast agent BR1; Sonazoid

STUDY DESIGN:
Intervention Model Description: included patients receive both SonoVue and Sonazoid with a randomized crossover design. The wash out period is at least 30min to make sure the fore-inject contrast agent is clear in blood.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The sequence of sonovue or sonazoid is blind to participant. The data is blind to the radiologist who is plan to evalutaed the data using CEUS LIRADS version 2017 and the outcome assessor who calculated all data and do the statistical calculation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonovue and Sonazoid Group (Experimental): Subjects were randomized to receive SonoVue firstly and Sonazid secondly after wash out period. Between the wash out period(at least 30min) and after whole trial, the patients was carefully observed at observing room for at least 30min.
  Contast agent dose: Sonazoid (0.12 μL/kg of perflubutane microbubbles) or SonoVue (2.4 mL) in a 1:1 ratio.
  Interventions: Drug: Sonovue and Sonazoid
- Sonazoid and Sonovue Group (Experimental): Subjects were randomized to receive Sonazoid firstly and SonoVue secondly after wash out period. Between the wash out period(at least 30min) and after whole trial, the patients was carefully observed at observing room for at least 30min.
  contast agent dose: Sonazoid (0.12 μL/kg of perflubutane microbubbles) or SonoVue (2.4 mL) in a 1:1 ratio.
  Interventions: Drug: Sonazoid and Sonovue

INTERVENTIONS:
Drug: Sonovue and Sonazoid — Subjects were randomized to receive SonoVue firstly and Sonazid secondly after wash out period. Between the wash out period(at least 30min) and after whole trial, the patients was carefully observed at our department for at least 30min.
  contast agent dose: Sonazoid (0.12 μL/kg of perflubutane microbubbles) or SonoVue (2.4 mL) in a 1:1 ratio.
  Arms: Sonovue and Sonazoid Group
Drug: Sonazoid and Sonovue — Subjects were randomized to receive Sonazoid firstly and SonoVue secondly after wash out period. Between the wash out period(at least 30min) and after whole trial, the patients was carefully observed at our department for at least 30min.
  contast agent dose: Sonazoid (0.12 μL/kg of perflubutane microbubbles) or SonoVue (2.4 mL) in a 1:1 ratio.
  Arms: Sonazoid and Sonovue Group

SUMMARY:
The new version of CEUS LI-RADS published at 2018(version 2017). In this study, the investigators aim to investigate the diagnosing performance of CEUS LI-RADS by administrating different contrast agents (SonoVue/ Sonazoid).

DETAILED DESCRIPTION:
Independent radiologists from department of ultrasound will report their diagnosing results according to CEUS LI-RADS version 2017 without getting any information about patients. The researcher of this subject will collect all results and evaluated the sensitivity and specificity of CEUS LI-RADS and the diagnosing performance with different contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk for HCC with focal liver lesion on conventional ultrasound.
* history of cirrhosis.
* historty of HBV infection.

Exclusion Criteria:

* systemic therapy with sorafenib
* pretreat lesion
* patients don't sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
CEUS LI-RADS Grades of SonoVue and Sonazoid agents in enrolled patients. | 6 months
  CEUS LI-RADS® v2017 which is published by ACR is a standardized system for technique, interpretation, reporting, and data collection for contrast-enhanced ultrasound exams in patients at risk for developing HCC.

SECONDARY OUTCOMES:
The sensitivity and specificity of CEUS-LI-RADS by different contrast agencies. | 6 months
  The sensitivity and specificity are calculated using parameters such as ture postive, false positive, Ture negative, false negetive.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ultrasound, The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China